CLINICAL TRIAL: NCT06246422
Title: The Effect of Local Instillation of Tranexamic Acid on the Gallbladder Bed After Laparoscopic Cholecystectomy to Decrease Possible Bleeding: Randomized Controlled Study.
Brief Title: Tranexamic Acid Instillation in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TXA/08/2022
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Complications
Keywords: gall bladder; postoperative bleeding; tranexamic acid
MeSH Terms: conditions — Postoperative Complications; Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants and the investigator will be kept blinded by the aid of closed sealed envelops. The measurements will be collected by the aid of assistant resident who will not participating into the study and blinded to it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): after careful hemostasis for the bleeding points in the liver bed received 500 mg of Tranexamic acid dissolved in 20 ml normal saline locally in the liver bed through the right port, then introduction of a piece of gauze to keep the drug in place for about 3 minutes and then remove it and inserting a drain and close it for one hour after finishing the operation.
  Interventions: Drug: Tranexamic Acid 500 MG
- group B (Experimental): they also underwent the same procedure with routine care for hemostasis until there was no significant bleeding and then instillation of 20 ml normal saline in the gallbladder bed , then drain was inserted and closed for 1 hour the sameway as group A.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Local instillation of 500 mg tranexamic acid in 20 ml normal saline in the gall bladder bed
  Arms: group A
Drug: Normal saline — Local instillation of 20 ml normal saline in the gall bladder bed
  Arms: group B

SUMMARY:
Adult patients undergoing laparoscopic cholecystectomy are at high risk to develop postoperative bleeding especially in the presence of severe adhesions. Local instillation of the antifibrinolytic (tranexamic acid) at the gall bladder bed may decrease the risk of bleeding.

The aim of this study is to evaluate the role of topical administration of Tranexamic acid on gallbladder bed for prophylaxis against bleeding in cases of difficult dissection cases due to acute inflammation and dense adhesions.

DETAILED DESCRIPTION:
This prospective study will be conducted in 80 adult patients admitted to surgery department Tanta University, the study will be carried out over 6 months after obtaining ethical committee approval, an informed written consent will be included.

Any unexpected risk that will appear during the procedure will be announced to the participants and ethical committee at time and adequate measures will be taken.

Risk to the patients There is known risk to the patient except for rare possible allergy to the drug.

All participant surgeons are experienced and familiar with the field. There will be adequate supervision to maintain the privacy of patients and confidentiality.

There will be no conflict of interest nor conflict with religion, law or society standards.

End point of study This study will be terminated if there is any unexpected risk from the drug.

This is a prospective study performed on 80 patients suffering from symptomatic cholelithiasis and will undergo laparoscopic cholecystectomy, they will be divided into two groups randomly by slip method. And will be performed by experienced surgeons.

All patients were subjected to:

Detailed history including drug intake (anticoagulants or antiplatelets) and thorough clinical examination.

laboratory investigations complete blood count (CBC), C-reactive protein (CRP), fasting blood sugar, renal function tests, and abdominal ultrasonography done.

Operative procedure After applying general anaesthesia , standard 4 port laparoscopic cholecystectomy will be performed. Patients in group A (40 patients) will receive 500 mg of Tranexamic acid dissolved in 20 ml normal saline locally in the liver bed after completing the procedure, we will introduce a piece of gauze to keep the drug in place for about 3 minutes and then remove it and we will insert a drain and close it for one hour after finishing the operation, if there is easy going operation without any adhesions and very minimal risk for bleeding it will be excluded.

For group B (40 patients) they will also undergo the same procedure with routine care that there is no significant bleeding then instillation of 20 ml normal saline locally in the liver bed and introduce a piece of gauze to keep the drug in place for about 3 minutes and then remove it and drain will be inserted for difficult cases and also easy ones will be excluded.

Post operative care Heart rate and blood pressure will be checked every 6 hours after surgery. Drain output will be recorded drain fluid hematocrit and hemoglobin will be investigated after 6 hours and 24 hours, and all the patients will be followed up till discharged. Drain will be removed if less than 50 cc for 24 hours.

Hb level will be performed after 48 h and was compared with the preoperative levels.

Any possible morbidity and time for ambulation and hospital stay will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21-60 years that underwent laparoscopic cholecystectomy with intra-operative difficult dissection due to adhesions or acute inflammation.

Exclusion Criteria:

* Patients who will refuse participation in the study
* Patients with bleeding disorders, clotting abnormalities, or on anticoagulants therapy.
* Easy going operation that do not necessitate drain insertion.
* major bleeding that could necessitate surgical intervention to control.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Hematocrit concentration in the drain | 6 hours
  The level of hematocrit in the drain 6 h after surgery

SECONDARY OUTCOMES:
Hemoglobin level in the drain | 6 hours
  The hemoglobin concentration in the drain 6 h after surgery
Length of hospital stay. | 24 hours
  Time from admission to discharge of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Once the study had been successfully completed, the data will be shared for other research